CLINICAL TRIAL: NCT06701513
Title: Registry of Psoriasis Health Outcomes: A Longitudinal Real-world Collaboration (RePhlect) - A Real-world, Prospective, Observational Study of the Effectiveness of Deucravacitinib in Adults With Moderate-to-Severe Plaque Psoriasis in France
Brief Title: A Real-world Study to Evaluate the Effectiveness of Deucravacitinib in Adults With Plaque Psoriasis in France (RePhlect)
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM011-1127
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — deucravacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Participants that have initiated deucravacitinib treatment
  Interventions: Drug: Deucravacitinib

INTERVENTIONS:
Drug: Deucravacitinib — As prescribed by treating clinician

SUMMARY:
The purpose of this study is to assess the real-world effectiveness of deucravacitinib treatment in adults diagnosed with moderate-to-severe plaque psoriasis

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Physician-reported diagnosis of moderate to severe plaque psoriasis
* Be newly initiating deucravacitinib
* Do not object to participate

Exclusion Criteria:

* Currently participating in or planning to participate in an interventional clinical trial
* Previous treatment experience with deucravacitinib, including patients who received deucravacitinib as part of a blinded, randomized trial

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients who have been diagnosed with moderate-to-severe plaque psoriasis and who intend to start deucravacitinib treatment in France
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Physician's Global Assessment (PGA) 0/1 response | Baseline and at months 4, 12, 18 (optional), and 24
Dermatology Life Quality Index (DLQI) 0/1 response | Baseline and at months 4, 12, 18 (optional), and 24
Time from date of treatment initiation to date of discontinuation | Up to 24 months

SECONDARY OUTCOMES:
Change in percentage involved Body Surface Area (BSA) from start of deucravacitinib treatment | Baseline and at months 4, 12, 18 (optional), and 24
Change in patient reported symptom burden as assed by the 100-point Visual Analog Scale (VAS) - Itch | Baseline and months 1, 4, 12, 18 (optional) and 24
Change in patient reported symptom burden as assed by the 100-point Visual Analog Scale (VAS) - Skin pain | Baseline and months 1, 4, 12, 18 (optional) and 24
Change in patient reported symptom burden as assed by the 100-point Visual Analog Scale (VAS)] - Fatigue | Baseline and months 1, 4, 12, 18 (optional) and 24
Physician's Global Assessment (PGA) score change from start of deucravacitinib treatment to follow-up | Baseline and at months 4, 12, 18 (optional), and 24
Dermatology Life Quality Index (DLQI) score of ≤5 | Baseline and at months 1, 4, 12 18 (optional) and 24
Body Surface Area (BSA) of ≤ 3% | Baseline and at months 4, 12, 18 (optional), and 24
Body Surface Area (BSA) of ≤ 1% | Baseline and at months 4, 12, 18 (optional), and 24
Reasons for deucravacitinib treatment discontinuation | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (39):
- France (33):
  - Local Institution - 060, Amiens
  - Cabinet Médical Elisabeth Lion, Angers
  - Local Institution - 045, Argenteuil
  - CH ARRAS, Arras
  - Local Institution - 041, Bordeaux
  - Local Institution - 048, Bordeaux
  - Centre Hospitalier William Morey - Hématologie, Chalon-sur-Saône
  - CHU Dijon, Dijon
  - Local Institution - 077, Dijon
  - Local Institution - 011, La Tronche
  - Local Institution - 074, Le Puy-en-Velay
  - Local Institution - 039, Lens
  - Local Institution - 004, Marcq-en-Barœul
  - Local Institution - 036, Montpellier
  - Local Institution - 012, Nice
  - Local Institution - 008, Niort
  - Local Institution - 070, Niort
  - Local Institution - 062, Nîmes
  - Local Institution - 073, Paris
  - Local Institution - 078, Périgueux
  - Local Institution - 046, Roubaix
  - Local Institution - 047, Roubaix
  - Local Institution - 051, Saint-Mandé
  - Local Institution - 072, Saint-Maur-des-Fossés
  - Hia Sainte Anne, Toulon
  - Local Institution - 054, Toulon
  - Local Institution - 005, Toulouse
  - Local Institution - 021, Toulouse
  - Local Institution - 037, Toulouse
  - Local Institution - 061, Vandœuvre-lès-Nancy
  - Local Institution - 064, Vandœuvre-lès-Nancy
  - Local Institution - 003, Villeurbanne
  - Local Institution - 006, Villeurbanne
- Switzerland (6):
  - Cabinet Medical, La Chaux-de-Fonds
  - Local Institution - 007, La Chaux-de-Fonds
  - Local Institution - 025, La Chaux-de-Fonds
  - Local Institution - 029, La Chaux-de-Fonds
  - Local Institution - 038, La Chaux-de-Fonds
  - Local Institution - 044, La Chaux-de-Fonds

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts